CLINICAL TRIAL: NCT03091972
Title: Left Atrial Liner Block Using Contact-force Catheter in Ablation for Atrial Fibrillation
Brief Title: Liner Ablation Using Contact-force in Atrial Fibrillation
Acronym: LIBCAAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Young-Hoon Kim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIBCAAF study
Record Dates: First submitted 2017-01-31; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Linear ablation; Catheter ablation; Contact force
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contact force assisted linear ablation (Experimental): Left atrial linear ablation performed using the contact force sensing catheter after pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Contact force assisted left atrial linear ablation
- control (Active Comparator): Left atrial linear ablation performed using the catheter without contact force sensing after pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation; Procedure: left atrial linear ablation without contact force monitoring

INTERVENTIONS:
Procedure: Pulmonary vein isolation — A pulmonary vein isolation procedure will be performed using radiofrequency ablation with contact force monitoring.
Procedure: Contact force assisted left atrial linear ablation — Left atrial linear ablation (Roof line and Anterior line) after pulmonary vein isolation during catheter ablation for persistent atrial fibrillation monitoring contact force.
  Arms: Contact force assisted linear ablation
Procedure: left atrial linear ablation without contact force monitoring — Left atrial linear ablation (Roof line and Anterior line) after pulmonary vein isolation during catheter ablation for persistent atrial fibrillation without monitoring contact force.
  Arms: control

SUMMARY:
Linear ablation is frequently used in the procedure for persistent atrial fibrillation. However, it has a limitation because of technical difficulty. Incomplete block is common and an important cause of atrial tachycardia.

The association between contact force values and successful linear block has not been revealed yet. We aim to the effectiveness and safety of linear ablation by using CF sensing catheter.

DETAILED DESCRIPTION:
Catheter ablation is currently accepted as a treatment option for symptomatic atrial fibrillation. Linear ablation is frequently used in the procedure for persistent atrial fibrillation. Multiple studies have shown benefit of linear ablation. However, it has a limitation because of technical difficulty. Incomplete block is common and an important cause of atrial tachycardia.

Contact-force (CF) monitoring during procedure has recently been available. This technology appears to significantly decrease procedure time and short term reconnection incidence in pulmonary vein (PV) isolation. It also helped to resolve the cause of PV reconnection. Some reports demonstrated that the association between reconnection and lower CF value.

Linear ablation has more variation to interrupt block and reconnection was more often than PV isolation. The association between CF values and successful linear block has not been revealed yet. In addition, the investigators aim to the effectiveness and safety of linear ablation by using CF sensing catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is18 years or greater
* Patients with persistent AF (AF episode lasting > 7 days)
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication
* Patients with recurrent or sustained arrhythmia after pulmonary vein isolation
* Patients undergoing a first-time ablation procedure for AF
* At least one episode of AF must have been documented by ECG, Holter, loop recorder, telemetry, trans telephonic monitoring (TTM), or implantable device within last 2 years of enrollment in this investigation
* Patients must be able and willing to provide written informed consent to participate in this investigation

Exclusion Criteria:

* Patients with long-standing persistent AF;
* Long-standing persistent AF will be defined as a sustained episode lasting more than 3 years.
* Patients for whom cardioversion or sinus rhythm will never be attempted/pursued;
* Patients with AF felt to be secondary to an obvious reversible cause
* Patients with contraindications to systemic anticoagulation with heparin or warfarin or a direct thrombin inhibitor;
* Patients with left atrial size ≥ 60 mm (2D echocardiography, parasternal long axis view)
* Moderate to severe valvular disease
* Reduced left ventricular function (ejection fraction <40%)
* Patients who are pregnant. Pregnancy will be assessed by patients informing the physicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation/atrial tachycardia | 12 months
  Freedom from any documented episode of atrial fibrillation/atrial tachycardia occurring after a single ablation procedure and lasting longer than 30 seconds with/without antiarrhythmic medication

SECONDARY OUTCOMES:
Total radiofrequency energy | 12 months
  Total radiofrequency energy to achieve bidirectional block of linear lesion in left atrium
Total force value | 12 months
  Total force value for complete block of linear lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Medical Center Anam hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Fassini G, Riva S, Chiodelli R, Trevisi N, Berti M, Carbucicchio C, Maccabelli G, Giraldi F, Bella PD. Left mitral isthmus ablation associated with PV Isolation: long-term results of a prospective randomized study. J Cardiovasc Electrophysiol. 2005 Nov;16(11):1150-6. doi: 10.1111/j.1540-8167.2005.50192.x. PMID 16302895
- [Result] Hocini M, Jais P, Sanders P, Takahashi Y, Rotter M, Rostock T, Hsu LF, Sacher F, Reuter S, Clementy J, Haissaguerre M. Techniques, evaluation, and consequences of linear block at the left atrial roof in paroxysmal atrial fibrillation: a prospective randomized study. Circulation. 2005 Dec 13;112(24):3688-96. doi: 10.1161/CIRCULATIONAHA.105.541052. PMID 16344401
- [Result] Willems S, Klemm H, Rostock T, Brandstrup B, Ventura R, Steven D, Risius T, Lutomsky B, Meinertz T. Substrate modification combined with pulmonary vein isolation improves outcome of catheter ablation in patients with persistent atrial fibrillation: a prospective randomized comparison. Eur Heart J. 2006 Dec;27(23):2871-8. doi: 10.1093/eurheartj/ehl093. Epub 2006 Jun 16. PMID 16782716
- [Result] Gaita F, Caponi D, Scaglione M, Montefusco A, Corleto A, Di Monte F, Coin D, Di Donna P, Giustetto C. Long-term clinical results of 2 different ablation strategies in patients with paroxysmal and persistent atrial fibrillation. Circ Arrhythm Electrophysiol. 2008 Oct;1(4):269-75. doi: 10.1161/CIRCEP.108.774885. PMID 19808418
- [Result] Santucci PA. Linear ablation of atrial fibrillation: what does it do? Heart Rhythm. 2010 Dec;7(12):1738-9. doi: 10.1016/j.hrthm.2010.09.001. Epub 2010 Sep 28. No abstract available. PMID 20817018
- [Result] Kautzner J, Neuzil P, Lambert H, Peichl P, Petru J, Cihak R, Skoda J, Wichterle D, Wissner E, Yulzari A, Kuck KH. EFFICAS II: optimization of catheter contact force improves outcome of pulmonary vein isolation for paroxysmal atrial fibrillation. Europace. 2015 Aug;17(8):1229-35. doi: 10.1093/europace/euv057. Epub 2015 Jun 3. PMID 26041872
- [Result] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733
- [Result] Andreu D, Gomez-Pulido F, Calvo M, Carlosena-Remirez A, Bisbal F, Borras R, Benito E, Guasch E, Prat-Gonzalez S, Perea RJ, Brugada J, Berruezo A, Mont L. Contact force threshold for permanent lesion formation in atrial fibrillation ablation: A cardiac magnetic resonance-based study to detect ablation gaps. Heart Rhythm. 2016 Jan;13(1):37-45. doi: 10.1016/j.hrthm.2015.08.010. Epub 2015 Aug 10. PMID 26272524
- [Result] le Polain de Waroux JB, Weerasooriya R, Anvardeen K, Barbraud C, Marchandise S, De Meester C, Goesaert C, Reis I, Scavee C. Low contact force and force-time integral predict early recovery and dormant conduction revealed by adenosine after pulmonary vein isolation. Europace. 2015 Jun;17(6):877-83. doi: 10.1093/europace/euu329. Epub 2015 Jan 24. PMID 25618742